CLINICAL TRIAL: NCT00600210
Title: AVF3963s Neoadjuvant Bevacizumab and Carboplatin Followed by Concurrent Bevacizumab, Carboplatin and Radiotherapy in the Primary Treatment of Cervix Cancer
Brief Title: Neoadjuvant Bevacizumab and Carboplatin Followed by Concurrent Bevacizumab, Carboplatin and Radiotherapy in the Primary Treatment of Cervix Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: low patient accrual
Sponsor: Leo W. Jenkins Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVF3963s
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Bevacizumab; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be delivered intravenously on day -7 at a dose of 10 mg/kg followed by carboplatin AUC 2.0 intravenously. This will allow therapy to start one week before starting radiotherapy to assess the initial tolerability of the combination without having radiation as a confounding factor, to start treatment while the patient's radiation is being planned, and to possibly optimize the tumor vasculature and allow optimal carboplatin delivery by the time chemoradiotherapy starts. Thereafter, bevacizumab will be given intravenously at 10 mg/kg every two weeks. Carboplatin will be given intravenously weekly at AUC 2.0. On weeks where both drugs are given, bevacizumab will be given first since it could help sensitize the tumor cells to carboplatin.
Drug: Carboplatin — Bevacizumab will be delivered intravenously on day -7 at a dose of 10 mg/kg followed by carboplatin AUC 2.0 intravenously. This will allow therapy to start one week before starting radiotherapy to assess the initial tolerability of the combination without having radiation as a confounding factor, to start treatment while the patient's radiation is being planned, and to possibly optimize the tumor vasculature and allow optimal carboplatin delivery by the time chemoradiotherapy starts. Thereafter, bevacizumab will be given intravenously at 10 mg/kg every two weeks. Carboplatin will be given intravenously weekly at AUC 2.0. On weeks where both drugs are given, bevacizumab will be given first since it could help sensitize the tumor cells to carboplatin.
Radiation: Radiation Therapy — Whole pelvis will be treated to a total dose of 45 Gy in 5 weeks.
  Cesium will be used with standard intracavitary systems preferably in two intracavitary applications. An effort should be made to deliver a minimum cumulative external and intracavitary dose to Point A of 85 Gy in 2 insertions.

SUMMARY:
This trial is designed to study the safety and efficacy of the combination of carboplatin, bevacizumab, and pelvic radiation therapy.

Rationale for substituting cisplatin with carboplatin:

Five landmark trials in cervical cancer prompted the National Cancer Institute in February of 1999 to issue a clinical announcement stating that "strong consideration should be given to adding concurrent chemotherapy in the treatment of invasive cervical cancer". The chemotherapeutic agent which was a common denominator to all 5 trials was cisplatin, and ever since it has become part of the standard of care for the treatment of stage IIB, III, and IVA cervical cancers. In addition, chemoradiotherapy with cisplatin is also considered one of the standard treatment options for IB2 and IIA tumors greater than 4 cm in diameter.

The most recent Gynecologic Oncology Group protocols for cervical cancer have used cisplatin and radiation therapy as in two of the five landmark trials. However, the benefit in survival given by cisplatin has not been without toxicity. In summary, in the trial by Keys 35% of patients receiving cisplatin and radiotherapy experienced moderate or severe toxicities. In the one by Rose, only 49 % completed the intended 6 cycles of chemotherapy.

Based on the toxicity profile of cisplatin, Higgins performed a phase II study of concurrent carboplatin with pelvic radiation therapy in the primary treatment of cervix cancer. He demonstrated the ability to administer carboplatin with concurrent radiation therapy with significantly less toxicity and with 94 % of the planned treatments delivered.

A comprehensive analysis of the literature from 1998 which compared the efficacy of carboplatin versus cisplatin in solid tumors concluded that for ovarian cancer and lung cancer the effectiveness of carboplatin was comparable to cisplatin, while for germ cell tumors, bladder cancer, and head and neck cancer cisplatin appeared superior. There was no mention of cervical cancer in this review, since at present there is no phase III trial comparing carboplatin versus cisplatin in cervix cancer.

Rationale for bevacizumab:

Bevacizumab is a recombinant humanized monoclonal IgG1 antibody that binds to and inhibits the biologic activity of vascular endothelial growth factor (VEGF) which stimulates tumor and tumor blood vessel growth. Targeting VEGF with bevacizumab could potentially be of benefit in cervical cancer patients by starving the tumor's blood supply and potentially enhancing the effect of radiotherapy and carboplatin chemotherapy.

DETAILED DESCRIPTION:
Five landmark trials in cervical cancer prompted the National Cancer Institute in February of 1999 to issue a clinical announcement stating that "strong consideration should be given to adding concurrent chemotherapy in the treatment of invasive cervical cancer". The chemotherapeutic agent which was a common denominator to all 5 trials was cisplatin, and ever since it has become part of the standard of care for the treatment of stage IIB, III, and IVA cervical cancers. In addition, chemoradiotherapy with cisplatin is also considered one of the standard treatment options for IB2 and IIA tumors greater than 4 cm in diameter.

The most recent GOG protocols for cervical cancer have used cisplatin 40 mg/m2 on days 1, 8, 15, 22, 29 of radiation therapy and once during parametrial brachytherapy boost for a total of 6 cycles. This cisplatin schedule was used in 2 of the 5 landmark trials by Rose [3] and Keys [4], respectively. However, the benefit in survival given by cisplatin, has not been without toxicity. Note that in the trial reported by Rose there was no radiotherapy alone arm for comparison. In summary, in the trial by Keys 35% of patients experienced grade 3 (moderate) or grade 4 (severe) toxicities, compared with 13 % in the radiotherapy alone arm. Specifically, 21 % experienced grade 3 or 4 leukopenia. Similarly, in the one by Rose, 23 % experienced grade 3 or 4 leukopenia, and only 49.4 % completed the intended 6 cycles of chemotherapy.

Based on the toxicity profile of cisplatin, Higgins et al. [5] performed a phase II study of concurrent carboplatin with pelvic radiation therapy in the primary treatment of cervix cancer. They demonstrated the ability to administer carboplatin dose based on an AUC of 2.0 on schedule with concurrent radiation therapy in the treatment of cervix cancer. Grade 3 leukopenia was observed in only 10 % of the patients, and no grade 4 leukopenia was observed. This is approximately half the incidence of leukopenia seen with cisplatin. More importantly, carboplatin was administered with an AUC of 2 in 175 out of 186 (94%) planned treatments. Treatment with carboplatin in this study had a similar excellent response rate, but with reduced hematologic side effects. A comprehensive analysis of the literature from 1998 which compared the efficacy of carboplatin versus cisplatin in solid tumors concluded that for ovarian cancer and lung cancer the effectiveness of carboplatin was comparable to cisplatin, while for germ cell tumors, bladder cancer, and head and neck cancer cisplatin appeared superior [6]. There was no mention of cervical cancer in this review, since at present there is no phase III trial comparing carboplatin versus cisplatin in cervix cancer.

Targeted therapies

Angiogenesis has been described in the majority of the cancer types affecting the female genital tract [7-14]. Multiple growth factors and cytokines are involved in the angiogenic process that accompanies cervical carcinogenesis. VEGF has a predominant role acting as an endothelial cell specific mitogen [15-17], and stimulates cell proliferation and increases vascular permeability. Various cancer types including breast, endometrial, ovarian, bladder, and lung cancer exhibit elevated VEGF expression at advanced stages [18-25], and has also been associated with high-grade intraepithelial lesions and cervical cancer [26-32]. VEGF protein levels have been shown to correlate with local tumor progression, metastasis and poor prognosis in the uterine cervix, based on immunohistochemical or enzyme immunoassay studies [26-31]. In patients undergoing primary radiotherapy for cervical cancer, serum VEGF influenced the progression free survival [33]. However, other reports have suggested that VEGF does not have a prognostic value [32]. In addition, Soufla et al. found a highly significant increase of VEGF mRNA expression upon cervical neoplastic transformation, and that high-grade squamous intraepithelial lesions exhibited higher VEGF mRNA levels than low-grade lesions [34].

Treatment of endothelial cells with carboplatin significantly increases the expression of VEGF [35]. Neutralization of secreted VEGF with specific polyclonal anti-VEGF antibodies sensitizes endothelial cells to carboplatin treatment and increases apoptosis several-fold [35]. Treatment with polyclonal anti-VEGF antibodies and carboplatin has been shown in vivo models to significantly enhance solid tumor growth inhibition over individual monotherapies [35]. Therefore, targeting VEGF could potentially be of benefit in cervical cancer patients.

Bevacizumab is a recombinant humanized monoclonal IgG1 antibody that binds to and inhibits the biologic activity of VEGF. Since bevacizumab may cause proteinuria and hypertension, carboplatin, which has less potential for renal toxicity than cisplatin, seems a better choice for combining with bevacizumab. The combination of radiotherapy, carboplatin, and bevacizumab could result in better results with decreased toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have IB2 and IIA tumors greater than 4 cm in diameter, IIB, IIIB without hydronephrosis or non-functioning kidney, and IVA without invasion to the bladder or rectum, primary, previously untreated, and histologically confirmed invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix.
* Negative, non-suspicious para-aortic nodes determined by CT lymphangiogram, MRI or lymphadenectomy.
* Adequate bone marrow function: ANC greater ≥ 1,500/mm3, platelets ≥ 100,000/mm3.
* Adequate renal function: serum creatinine ≤ 1.5 mg/100 mL.
* Adequate hepatic function: bilirubin less than or equal to 1.5 x upper limit of normal (ULN) and SGOT and alkaline phosphatase less than or equal to 3 x ULN.
* Zubrod Performance Status of 0 or 1
* Patients of childbearing potential must have a negative serum pregnancy test within14 days of enrolling in this study and use an effective form of contraception during the study period.
* Patients who are medically suitable for treatment with radical intent using concurrent chemotherapy and pelvic radiation.

Exclusion Criteria:

* Patients with Stage IA, IB1, IB2 and IIa tumors less than 4 cm in diameter, IIIA or IVB disease.
* Patients who have known metastases to para-aortic or scalene nodes or metastases to other organs outside the radiation field at the time of the original clinical and surgical staging.
* Extensive tumor preventing intracavitary irradiation.
* Distal vaginal involvement or any disease such that an interstitial implant might be necessary
* Previous pelvic or abdominal radiation, cytotoxic chemotherapy, or previous therapy of any kind for this malignancy.
* Patients who might require an emergency surgical procedure to relieve hydronephrosis, or who are at risk of perforating the bladder and might require surgery.
* Patients with renal abnormalities, such as pelvic kidney, horseshoe kidney, or renal transplantation, that would require modification of radiation fields
* Life expectancy of less than 12 weeks
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study.
* Septicemia or severe infection
* Patients who have circumstances that will not permit completion of this study or the required follow-up.
* Patients who are pregnant at the time of diagnosis and do not wish pregnancy termination prior to initiation of treatment.
* Other concomitant malignancies, with the exception of nonmelanoma skin cancer, who had (or have) any evidence of other cancer present within the last 5 years.
* Bevacizumab-Specific Exclusions
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Known CNS disease
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either
* Urine protein:creatinine (UPC) ratio ≥1.0 at screening OR
* Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab
* Pregnant (positive pregnancy test) or lactating. Use of effective means of contraception (men and women) in subjects of child-bearing potential
* Any history of stroke or transient ischemic attack at any time
* History of myocardial infarction or unstable angina within 6 months of study enrollment
* Carboplatin-Specific Exclusions
* History of severe allergic reactions to cisplatin or other platinum-containing compounds.
* Patients with severe bone marrow depression or significant bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety of the proposed treatment in this patient population. | 5 years

SECONDARY OUTCOMES:
Progression Free Survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Frelix, MD, Principal Investigator — East Carolina University School of Medicine
Locations (1):
- East Carolina University School of Medicine, Greenville, North Carolina, United States

REFERENCES:
- [Background] Jemal A, Murray T, Ward E, Samuels A, Tiwari RC, Ghafoor A, Feuer EJ, Thun MJ. Cancer statistics, 2005. CA Cancer J Clin. 2005 Jan-Feb;55(1):10-30. doi: 10.3322/canjclin.55.1.10. PMID 15661684
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Rose PG, Bundy BN, Watkins EB, Thigpen JT, Deppe G, Maiman MA, Clarke-Pearson DL, Insalaco S. Concurrent cisplatin-based radiotherapy and chemotherapy for locally advanced cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1144-53. doi: 10.1056/NEJM199904153401502. PMID 10202165
- [Background] Keys HM, Bundy BN, Stehman FB, Muderspach LI, Chafe WE, Suggs CL 3rd, Walker JL, Gersell D. Cisplatin, radiation, and adjuvant hysterectomy compared with radiation and adjuvant hysterectomy for bulky stage IB cervical carcinoma. N Engl J Med. 1999 Apr 15;340(15):1154-61. doi: 10.1056/NEJM199904153401503. PMID 10202166
- [Background] Higgins RV, Naumann WR, Hall JB, Haake M. Concurrent carboplatin with pelvic radiation therapy in the primary treatment of cervix cancer. Gynecol Oncol. 2003 Jun;89(3):499-503. doi: 10.1016/s0090-8258(03)00151-3. PMID 12798718
- [Background] Lokich J, Anderson N. Carboplatin versus cisplatin in solid tumors: an analysis of the literature. Ann Oncol. 1998 Jan;9(1):13-21. doi: 10.1023/a:1008215213739. PMID 9541678
- [Background] Abulafia O, Triest WE, Sherer DM. Angiogenesis in malignancies of the female genital tract. Gynecol Oncol. 1999 Feb;72(2):220-31. doi: 10.1006/gyno.1998.5152. PMID 10021305
- [Background] Tokumo K, Kodama J, Seki N, Nakanishi Y, Miyagi Y, Kamimura S, Yoshinouchi M, Okuda H, Kudo T. Different angiogenic pathways in human cervical cancers. Gynecol Oncol. 1998 Jan;68(1):38-44. doi: 10.1006/gyno.1997.4876. PMID 9454658
- [Background] Smith-McCune KK, Weidner N. Demonstration and characterization of the angiogenic properties of cervical dysplasia. Cancer Res. 1994 Feb 1;54(3):800-4. PMID 7508337
- [Background] Abulafia O, Triest WE, Sherer DM, Hansen CC, Ghezzi F. Angiogenesis in endometrial hyperplasia and stage I endometrial carcinoma. Obstet Gynecol. 1995 Oct;86(4 Pt 1):479-85. doi: 10.1016/0029-7844(95)00203-4. PMID 7545803
- [Background] Ishiwata I, Ishiwata C, Soma M, Ono I, Nakaguchi T, Ishikawa H. Tumor angiogenic activity of gynecologic tumor cell lines on the chorioallantoic membrane. Gynecol Oncol. 1988 Jan;29(1):87-93. doi: 10.1016/0090-8258(88)90151-5. PMID 2448191
- [Background] Abulafia O, Triest WE, Sherer DM. Angiogenesis in primary and metastatic epithelial ovarian carcinoma. Am J Obstet Gynecol. 1997 Sep;177(3):541-7. doi: 10.1016/s0002-9378(97)70143-1. PMID 9322621
- [Background] Nakanishi Y, Kodama J, Yoshinouchi M, Tokumo K, Kamimura S, Okuda H, Kudo T. The expression of vascular endothelial growth factor and transforming growth factor-beta associates with angiogenesis in epithelial ovarian cancer. Int J Gynecol Pathol. 1997 Jul;16(3):256-62. doi: 10.1097/00004347-199707000-00011. PMID 9421092
- [Background] Hollingsworth HC, Kohn EC, Steinberg SM, Rothenberg ML, Merino MJ. Tumor angiogenesis in advanced stage ovarian carcinoma. Am J Pathol. 1995 Jul;147(1):33-41. PMID 7541612
- [Background] Carmeliet P, Jain RK. Angiogenesis in cancer and other diseases. Nature. 2000 Sep 14;407(6801):249-57. doi: 10.1038/35025220. PMID 11001068
- [Background] Gasparini G. Clinical significance of determination of surrogate markers of angiogenesis in breast cancer. Crit Rev Oncol Hematol. 2001 Feb;37(2):97-114. doi: 10.1016/s1040-8428(00)00105-0. PMID 11166583
- [Background] Bergers G, Benjamin LE. Tumorigenesis and the angiogenic switch. Nat Rev Cancer. 2003 Jun;3(6):401-10. doi: 10.1038/nrc1093. PMID 12778130
- [Background] Brown LF, Berse B, Jackman RW, Tognazzi K, Guidi AJ, Dvorak HF, Senger DR, Connolly JL, Schnitt SJ. Expression of vascular permeability factor (vascular endothelial growth factor) and its receptors in breast cancer. Hum Pathol. 1995 Jan;26(1):86-91. doi: 10.1016/0046-8177(95)90119-1. PMID 7821921
- [Background] Boocock CA, Charnock-Jones DS, Sharkey AM, McLaren J, Barker PJ, Wright KA, Twentyman PR, Smith SK. Expression of vascular endothelial growth factor and its receptors flt and KDR in ovarian carcinoma. J Natl Cancer Inst. 1995 Apr 5;87(7):506-16. doi: 10.1093/jnci/87.7.506. PMID 7707437
- [Background] Abu-Jawdeh GM, Faix JD, Niloff J, Tognazzi K, Manseau E, Dvorak HF, Brown LF. Strong expression of vascular permeability factor (vascular endothelial growth factor) and its receptors in ovarian borderline and malignant neoplasms. Lab Invest. 1996 Jun;74(6):1105-15. PMID 8667614
- [Background] Xu L, Xie K, Mukaida N, Matsushima K, Fidler IJ. Hypoxia-induced elevation in interleukin-8 expression by human ovarian carcinoma cells. Cancer Res. 1999 Nov 15;59(22):5822-9. PMID 10582705
- [Background] Chen CA, Cheng WF, Lee CN, Chen TM, Kung CC, Hsieh FJ, Hsieh CY. Serum vascular endothelial growth factor in epithelial ovarian neoplasms: correlation with patient survival. Gynecol Oncol. 1999 Aug;74(2):235-40. doi: 10.1006/gyno.1999.5418. PMID 10419737
- [Background] Brown LF, Berse B, Jackman RW, Tognazzi K, Manseau EJ, Dvorak HF, Senger DR. Increased expression of vascular permeability factor (vascular endothelial growth factor) and its receptors in kidney and bladder carcinomas. Am J Pathol. 1993 Nov;143(5):1255-62. PMID 8238242
- [Background] Macchiarini P, Fontanini G, Hardin MJ, Squartini F, Angeletti CA. Relation of neovascularisation to metastasis of non-small-cell lung cancer. Lancet. 1992 Jul 18;340(8812):145-6. doi: 10.1016/0140-6736(92)93217-b. PMID 1378165
- [Background] Guidi AJ, Abu-Jawdeh G, Tognazzi K, Dvorak HF, Brown LF. Expression of vascular permeability factor (vascular endothelial growth factor) and its receptors in endometrial carcinoma. Cancer. 1996 Aug 1;78(3):454-60. doi: 10.1002/(SICI)1097-0142(19960801)78:33.0.CO;2-Y. PMID 8697391
- [Background] Guidi AJ, Abu-Jawdeh G, Berse B, Jackman RW, Tognazzi K, Dvorak HF, Brown LF. Vascular permeability factor (vascular endothelial growth factor) expression and angiogenesis in cervical neoplasia. J Natl Cancer Inst. 1995 Aug 16;87(16):1237-45. doi: 10.1093/jnci/87.16.1237. PMID 7563170
- [Background] Loncaster JA, Cooper RA, Logue JP, Davidson SE, Hunter RD, West CM. Vascular endothelial growth factor (VEGF) expression is a prognostic factor for radiotherapy outcome in advanced carcinoma of the cervix. Br J Cancer. 2000 Sep;83(5):620-5. doi: 10.1054/bjoc.2000.1319. PMID 10944602
- [Background] Lee IJ, Park KR, Lee KK, Song JS, Lee KG, Lee JY, Cha DS, Choi HI, Kim DH, Deung YK. Prognostic value of vascular endothelial growth factor in Stage IB carcinoma of the uterine cervix. Int J Radiat Oncol Biol Phys. 2002 Nov 1;54(3):768-79. doi: 10.1016/s0360-3016(02)02970-x. PMID 12377329
- [Background] Cheng WF, Chen CA, Lee CN, Chen TM, Hsieh FJ, Hsieh CY. Vascular endothelial growth factor in cervical carcinoma. Obstet Gynecol. 1999 May;93(5 Pt 1):761-5. doi: 10.1016/s0029-7844(98)00505-5. PMID 10912982
- [Background] Cheng WF, Chen CA, Lee CN, Wei LH, Hsieh FJ, Hsieh CY. Vascular endothelial growth factor and prognosis of cervical carcinoma. Obstet Gynecol. 2000 Nov;96(5 Pt 1):721-6. doi: 10.1016/s0029-7844(00)01025-5. PMID 11042307
- [Background] Gaffney DK, Haslam D, Tsodikov A, Hammond E, Seaman J, Holden J, Lee RJ, Zempolich K, Dodson M. Epidermal growth factor receptor (EGFR) and vascular endothelial growth factor (VEGF) negatively affect overall survival in carcinoma of the cervix treated with radiotherapy. Int J Radiat Oncol Biol Phys. 2003 Jul 15;56(4):922-8. doi: 10.1016/s0360-3016(03)00209-8. PMID 12829126
- [Background] Tjalma W, Weyler J, Weyn B, Van Marck E, Van Daele A, Van Dam P, Goovaerts G, Buytaert P. The association between vascular endothelial growth factor, microvessel density and clinicopathological features in invasive cervical cancer. Eur J Obstet Gynecol Reprod Biol. 2000 Oct;92(2):251-7. doi: 10.1016/s0301-2115(99)00295-x. PMID 10996690
- [Background] Bachtiary B, Selzer E, Knocke TH, Potter R, Obermair A. Serum VEGF levels in patients undergoing primary radiotherapy for cervical cancer: impact on progression-free survival. Cancer Lett. 2002 May 28;179(2):197-203. doi: 10.1016/s0304-3835(01)00872-2. PMID 11888674
- [Background] Soufla G, Sifakis S, Baritaki S, Zafiropoulos A, Koumantakis E, Spandidos DA. VEGF, FGF2, TGFB1 and TGFBR1 mRNA expression levels correlate with the malignant transformation of the uterine cervix. Cancer Lett. 2005 Apr 18;221(1):105-18. doi: 10.1016/j.canlet.2004.08.021. PMID 15797633
- [Background] Wild R, Dings RP, Subramanian I, Ramakrishnan S. Carboplatin selectively induces the VEGF stress response in endothelial cells: Potentiation of antitumor activity by combination treatment with antibody to VEGF. Int J Cancer. 2004 Jun 20;110(3):343-51. doi: 10.1002/ijc.20100. PMID 15095298
- [Background] Mathur RS, Mathur SP. Vascular endothelial growth factor (VEGF) up-regulates epidermal growth factor receptor (EGF-R) in cervical cancer in vitro: this action is mediated through HPV-E6 in HPV-positive cancers. Gynecol Oncol. 2005 Apr;97(1):206-13. doi: 10.1016/j.ygyno.2004.12.011. PMID 15790460
- [Background] Kristensen GB, Holm R, Abeler VM, Trope CG. Evaluation of the prognostic significance of cathepsin D, epidermal growth factor receptor, and c-erbB-2 in early cervical squamous cell carcinoma. An immunohistochemical study. Cancer. 1996 Aug 1;78(3):433-40. doi: 10.1002/(SICI)1097-0142(19960801)78:33.0.CO;2-K. PMID 8697388
- [Background] Kersemaekers AM, Fleuren GJ, Kenter GG, Van den Broek LJ, Uljee SM, Hermans J, Van de Vijver MJ. Oncogene alterations in carcinomas of the uterine cervix: overexpression of the epidermal growth factor receptor is associated with poor prognosis. Clin Cancer Res. 1999 Mar;5(3):577-86. PMID 10100709
- [Background] Cho NH, Kim YB, Park TK, Kim GE, Park K, Song KJ. P63 and EGFR as prognostic predictors in stage IIB radiation-treated cervical squamous cell carcinoma. Gynecol Oncol. 2003 Nov;91(2):346-53. doi: 10.1016/s0090-8258(03)00504-3. PMID 14599865
- [Background] Skomedal H, Kristensen GB, Lie AK, Holm R. Aberrant expression of the cell cycle associated proteins TP53, MDM2, p21, p27, cdk4, cyclin D1, RB, and EGFR in cervical carcinomas. Gynecol Oncol. 1999 May;73(2):223-8. doi: 10.1006/gyno.1999.5346. PMID 10329038
- [Background] Ngan HY, Cheung AN, Liu SS, Cheng DK, Ng TY, Wong LC. Abnormal expression of epidermal growth factor receptor and c-erbB2 in squamous cell carcinoma of the cervix: correlation with human papillomavirus and prognosis. Tumour Biol. 2001 May-Jun;22(3):176-83. doi: 10.1159/000050613. PMID 11275796
- [Background] Nagai N, Oshita T, Fujii T, Kioka H, Katsube Y, Ohama K. Prospective analysis of DNA ploidy, proliferative index and epidermal growth factor receptor as prognostic factors for pretreated uterine cancer. Oncol Rep. 2000 May-Jun;7(3):551-9. doi: 10.3892/or.7.3.551. PMID 10767367
- [Background] Scambia G, Ferrandina G, Distefano M, D'Agostino G, Benedetti-Panici P, Mancuso S. Epidermal growth factor receptor (EGFR) is not related to the prognosis of cervical cancer. Cancer Lett. 1998 Jan 30;123(2):135-9. doi: 10.1016/s0304-3835(97)00421-7. PMID 9489479
- [Background] Kim JW, Kim YT, Kim DK, Song CH, Lee JW. Expression of epidermal growth factor receptor in carcinoma of the cervix. Gynecol Oncol. 1996 Feb;60(2):283-7. doi: 10.1006/gyno.1996.0039. PMID 8631552
- [Background] Finlay MH, Ackerman I, Tirona RG, Hamilton P, Barbera L, Thomas G. Use of CT simulation for treatment of cervical cancer to assess the adequacy of lymph node coverage of conventional pelvic fields based on bony landmarks. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):205-9. doi: 10.1016/j.ijrobp.2005.06.025. Epub 2005 Sep 29. PMID 16198505
- [Background] Willett CG, Boucher Y, Duda DG, di Tomaso E, Munn LL, Tong RT, Kozin SV, Petit L, Jain RK, Chung DC, Sahani DV, Kalva SP, Cohen KS, Scadden DT, Fischman AJ, Clark JW, Ryan DP, Zhu AX, Blaszkowsky LS, Shellito PC, Mino-Kenudson M, Lauwers GY. Surrogate markers for antiangiogenic therapy and dose-limiting toxicities for bevacizumab with radiation and chemotherapy: continued experience of a phase I trial in rectal cancer patients. J Clin Oncol. 2005 Nov 1;23(31):8136-9. doi: 10.1200/JCO.2005.02.5635. No abstract available. PMID 16258121
- [Background] Kitayama H, Maeshima Y, Takazawa Y, Yamamoto Y, Wu Y, Ichinose K, Hirokoshi K, Sugiyama H, Yamasaki Y, Makino H. Regulation of angiogenic factors in angiotensin II infusion model in association with tubulointerstitial injuries. Am J Hypertens. 2006 Jul;19(7):718-27. doi: 10.1016/j.amjhyper.2005.09.022. PMID 16814127
- [Background] Lanciano R, Calkins A, Bundy BN, Parham G, Lucci JA 3rd, Moore DH, Monk BJ, O'Connor DM. Randomized comparison of weekly cisplatin or protracted venous infusion of fluorouracil in combination with pelvic radiation in advanced cervix cancer: a gynecologic oncology group study. J Clin Oncol. 2005 Nov 20;23(33):8289-95. doi: 10.1200/JCO.2004.00.0497. Epub 2005 Oct 17. PMID 16230678